CLINICAL TRIAL: NCT07041008
Title: Cognitive Stimulation in Older Adults With Alzheimer's Disease: Effects Across Multiple Domains and in Institutional and Sociogeographic Contexts
Brief Title: Cognitive Stimulation in Older Adults With Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rsocialform - Geriatria, Lda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13062025
Record Dates: First submitted 2025-06-17; First posted 2025-06-27 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Neurocognitive Disorders; Cognitive Impairment; Cognitive Dysfunction; Cognitive Decline
Keywords: older adults; cognitive function; memory; executive function; dementia; cognitive stimulation therapy; cognition; neurocognitive disorders; individual therapy; non-pharmacological therapy; mood; depression; anxiety; quality of life; randomised controlled trial; Alzheimer's disease
MeSH Terms: conditions — Dementia; Neurocognitive Disorders; Cognitive Dysfunction; Depression; Anxiety Disorders; Alzheimer Disease | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Experimental): Participants in the intervention group 1 will participate in two individual CS sessions per week for 12 weeks in addition to their treatment as usual. The sessions will include the same program in every participant site.
  Interventions: Behavioral: Digital intervention
- Intervention group 2 (Experimental): Participants in the intervention group 2 will participate in two individual CS sessions per week for 12 weeks in addition to their treatment as usual. The sessions will include the same program in every participant site.
  Interventions: Behavioral: Physical/Analogue Intervention
- Control group (No intervention) (No Intervention): Participants in the control group will receive treatment as usual (TAU) at the site, following the activities specified in their individual care plans.

INTERVENTIONS:
Behavioral: Digital intervention — Individual cognitive stimulation sessions will be delivered using RehaCom software, which provides adaptive, computerised exercises targeting specific cognitive domains.
  Arms: Intervention group 1
Behavioral: Physical/Analogue Intervention — Individual cognitive stimulation sessions will employ structured physical materials, specifically the 'Memories from North to South©' and 'Cognitive Domains' resources, applied on an alternating basis.
  Arms: Intervention group 2

SUMMARY:
This multicentre study, employing a randomised controlled repeated measures experimental design, will be conducted in several Portuguese institutions that provide care and support services for older adults diagnosed with mild to moderate Alzheimer's disease (AD). The primary aim is to evaluate the effects of two distinct cognitive stimulation modalities (digital vs physical/analogue).

The study will assess the impact of individual cognitive stimulation on multiple domains - specifically cognitive function (with an emphasis on memory and executive function), mood, and quality of life - and investigate how institutional and territorial characteristics influence these effects, considering geographical and organisational diversity as potential moderating factors.

DETAILED DESCRIPTION:
Population ageing has increased the prevalence of neurodegenerative diseases, with Alzheimer's disease (AD) being the most common form of dementia. Its wide-ranging impact on cognition, emotion, and daily function necessitates person-centred, multidimensional interventions. In Portugal, dementia affects around 9.5% of those aged 65+, underlining its public health relevance and the need for effective responses.

In the absence of a cure, non-pharmacological interventions like cognitive stimulation (CS) have gained prominence. CS is an evidence-based, psychosocial approach involving structured activities that enhance cognitive functions such as memory, language, attention, and reasoning. Broader and more relational than cognitive training or rehabilitation, CS is effective-especially in mild to moderate AD-in improving cognition, mood, and quality of life. Portuguese and international guidelines support its use, with studies showing potential in reducing depression and anxiety in older adults.

Behavioural and psychological symptoms of dementia (BPSD)-including agitation, apathy, aggression, anxiety, and sleep issues-are common in AD and often more disruptive than cognitive decline. These symptoms increase caregiver stress and the likelihood of institutionalisation. CS may alleviate BPSD through emotional engagement and behavioural regulation.

Assessing CS efficacy requires reliable tools. The Mini-Mental State Examination is widely used in Portugal for cognitive screening, while the Alzheimer's Disease Assessment Scale - Cognitive Subscale is often used in clinical trials. As AD notably impairs executive functions, CS targeting these domains can support autonomy and adaptive behaviour.

Contextual factors, such as institutional resources and geographic location, may influence CS outcomes. However, few studies consider these variables, despite their relevance for implementing sustainable, real-world interventions.

This research adopts a multicentre, randomised controlled design to examine two individual CS modalities in older adults with mild to moderate AD attending Portuguese social care services. It aims to assess CS effects on global cognition (particularly executive function and memory), mood, and quality of life, and to explore how institutional and territorial factors shape outcomes.

By combining validated measures, structured protocols, and a context-sensitive approach, the study seeks to support the implementation of effective, sustainable CS interventions within Portugal's care system.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older.
* Receive care/support services for at least three months.
* A diagnosis of probable AD according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, fifth edition, text revision.
* Preserved communication skills.
* Native Portuguese speaker.
* Total scores between 10 and 26 points on the Mini Mental State Examination.

Exclusion Criteria:

* Cannot read and write.
* Significant sensory or physical limitations.
* Acute or chronic illness preventing participation.
* Severe communication impairment.
* Aggressive or disruptive behaviour.
* Recent initiation (within two months) of neuroleptics, antipsychotics, or other psychoactive medications.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive functioning assessed through Mini-Mental State Examination (MMSE) | Baseline
  Cognitive functioning assessed by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning assessed through Mini-Mental State Examination (MMSE) | 12 weeks after the baseline
  Change in cognitive functioning evaluated by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function.Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning assessed through Mini-Mental State Examination (MMSE) | 24 weeks after the baseline
  Change in cognitive functioning evaluated by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | Baseline
  Evaluates the severity of cognitive deficits in AD in the following domains: memory, orientation, language, praxis and constructive capacity. The total score in the Portuguese version of ADAS-Cog is composed of 11 subtests in the cognitive part and varies between 0 (better performance) and 68 points (worse performance), i.e., higher scores equals better performance.
Change in cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | 12 weeks after the baseline
  Evaluates the severity of cognitive deficits in AD in the following domains: memory, orientation, language, praxis and constructive capacity. The total score in the Portuguese version of ADAS-Cog is composed of 11 subtests in the cognitive part and varies between 0 (better performance) and 68 points (worse performance), i.e., higher scores equals better performance.
Change in cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | 24 weeks after the baseline
  Evaluates the severity of cognitive deficits in AD in the following domains: memory, orientation, language, praxis and constructive capacity. The total score in the Portuguese version of ADAS-Cog is composed of 11 subtests in the cognitive part and varies between 0 (better performance) and 68 points (worse performance), i.e., higher scores equals better performance.
Memory function evaluated through Memory Alteration Test (MAT) | Baseline
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.
Change in memory function evaluated through Memory Alteration Test (MAT) | 12 weeks after the baseline
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.
Change in memory function evaluated through Memory Alteration Test (MAT) | 24 weeks after the baseline
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.
Executive functions assessed through Frontal Assessment Battery (FAB) | Baseline
  FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points with higher scores indicating better cognitive function.
Change in executive functions assessed through Frontal Assessment Battery (FAB) | 12 weeks after the baseline
  FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points with higher scores indicating better cognitive function.
Change in executive functions assessed through Frontal Assessment Battery (FAB) | 24 weeks after the baseline
  FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points with higher scores indicating better cognitive function.

SECONDARY OUTCOMES:
Mood assessed through the Geriatric Depression Scale-15 (GDS-15) | Baseline
  The GDS-15 is used to measure mood. It is considered a reliable tool to screen depressive symptoms in older people. With a dichotomous format (yes/no answers), this scale assesses depression in older people. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
Change in mood assessed through the GDS-15 | 12 weeks after the baseline
  The GDS-15 is used to measure mood. It is considered a reliable tool to screen depressive symptoms in older people. With a dichotomous format (yes/no answers), this scale assesses depression in older people. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
Change in mood assessed through the GDS-15 | 24 weeks after the baseline
  The GDS-15 is used to measure mood. It is considered a reliable tool to screen depressive symptoms in older people. With a dichotomous format (yes/no answers), this scale assesses depression in older people. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
Anxiety symptomatology assessed through the Geriatric Anxiety Inventory (GAI) | Baseline
  It assesses, in several contexts, the severity of anxiety symptoms in the older adults. It consists in 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Change in anxiety symptomatology assessed through the GAI | 12 weeks after the baseline
  It assesses, in several contexts, the severity of anxiety symptoms in the older adults. It consists in 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Change in anxiety symptomatology assessed through the GAI | 24 weeks after the baseline
  It assesses, in several contexts, the severity of anxiety symptoms in the older adults. It consists in 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Quality of life evaluated through Quality of Life - Alzheimer's Disease (QoL-AD) | Baseline
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.
Change in quality of life evaluated through QoL-AD | 12 weeks after the baseline
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.
Change in quality of life evaluated through QoL-AD | 24 weeks after the baseline
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life. It has good psychometric characteristics and its use has been recommended to evaluate psychosocial interventions.

OTHER OUTCOMES:
Sociodemographic, geographical and social information collected through the Sociodemographic, Geographical and Social Characteristics Questionnaire | Baseline
  Participants' responses to the Sociodemographic, Geographical and Social Characteristics Questionnaire, developed specifically for this study, will be collected. This questionnaire gathers data such as age, place of birth, gender, marital status, educational level, clinical condition, and pharmacological drugs. Additionally, relevant institutional and territorial variables will be recorded, including the geographical location of the institution (urban, rural, or mixed area), type and legal status of the social service, number of users, availability of rooms and equipment suitable for the intervention, and training of the cognitive stimulation team. The questionnaire will be administered to all participants.
Adherence to the intervention and dropouts evaluated through a session form | up to 12 weeks after baseline
  Adherence to the intervention and dropouts will be assessed using a session form, designed specifically for this study, completed by the technician after each session, regarding the attendance and mood/behavior of the participants throughout the intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I. Justo Henriques, PhD, Principal Investigator — Polytechnic University of Beja
Locations (39):
- Portugal (39):
  - AMITEI, Leiria, Leria
  - Associação de Desenvolvimento Comunitário do Funchal - Garouta do Calhau, Funchal, Madeira
  - Instituto S. João de Deus Funchal, Funchal, Madeira
  - Associação Alzheimer Açores, Açores
  - Santa Casa da Misericórdia da Horta, Açores
  - Santa Casa da Misericórdia de Vila do Porto, Açores
  - CASTIIS, Aveiro
  - CEDIARA - Associação de Solidariedade Social de Ribeira de Fráguas, Aveiro
  - Centro Apoio Social Mozelos, Aveiro
  - Centro Social da Freguesia de Casal Comba, Aveiro
  - O Jardim - Centro de Solidariedade Social de Canedo, Aveiro
  - Santa Casa da Misericórdia de Espinho, Aveiro
  - Santa Casa da Misericórdia de Ovar, Aveiro
  - Patronato de Santo António - Lar D. José do Patrocínio Dias, Beja
  - Santa Casa da Misericórdia de Ferreira do Alentejo, Beja
  - Centro Social do Vale do Homem Casa da Alegria, Braga
  - Santa Casa da Misericórdia de Mirandela, Bragança
  - Residência Sénior DON ANTÓNIO - Hilário & Pereira, Castelo Branco
  - Santa Casa da Misericórdia da Soalheira, Castelo Branco
  - Santa Casa da Misericórdia de Vila Velha de Rodão, Castelo Branco
  - Associação Cultural Recreativa e Social de Samuel, Coimbra
  - Santa Casa da Misericórdia de Montemor-o-Novo, Evora
  - Santa Casa da Misericórdia de Vila Real de Santo António, Faro
  - Fundação João Bento Raimundo, Guarda
  - Santa Casa da Misericórdia de Figueira de Castelo Rodrigo, Guarda
  - Santa Casa da Misericórdia de Alcobaça, Leiria
  - Santa Casa da Misericórdia de Alvaiázere, Leiria
  - Santa Casa da Misericórdia de Alvorge, Leiria
  - Associação Casapiana de Solidariedade, Lisbon
  - Associação de Socorros da Freguesia de Turcifal, Lisbon
  - Centro Social Paroquial de Moita dos Ferreiros, Lisbon
  - Santa Casa da Misericórdia de Lisboa - Espaço ComVida, Lisbon
  - Santa Casa da Misericórdia de Campo Maior, Portalegre
  - Santa Casa da Misericórdia de Gaia - ERPI José Tavares Bastos, Porto
  - Quinta de Santa Ana RS, Viana do Castelo
  - Santa Casa da Misericórdia de Caminha, Viana do Castelo
  - Santa Casa da Misericórdia de Ponte de Lima, Viana do Castelo
  - Associação de Solidariedade Social do Alto Paiva, Viseu
  - Associação de Solidariedade Social e Recreativa de Nespereira, Viseu

IPD SHARING:
Plan to Share IPD: No